CLINICAL TRIAL: NCT06333808
Title: Phase 3 Double-blind Multicenter Randomized Active-Controlled Study to Evaluate the Safety and Efficacy of Bictegravir/Lenacapavir Versus Biktarvy® (Bictegravir/Emtricitabine/Tenofovir Alafenamide) in Virologically Suppressed People With HIV-1
Brief Title: Study to Compare Bictegravir/Lenacapavir Versus Current Therapy in People With HIV-1 Who Are Successfully Treated With Biktarvy
Acronym: ARTISTRY-2
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GS-US-621-6290; 2023-510022-33 (Other: European Medicines Agency); jRCT2051240046 (Registry Identifier: Japan Registry)
Record Dates: First submitted 2024-03-20; First posted 2024-03-27 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-11

CONDITIONS: HIV-1-infection
MeSH Terms: interventions — bictegravir; lenacapavir; bictegravir, emtricitabine, tenofovir alafenamide, drug combination

STUDY DESIGN:
Intervention Model Description: Participants will be randomized in parallel in one of two treatment groups during the Blinded Phase. Participants in both treatment groups will be given the option to continue BIC/LEN FDC treatment during the Open-Label Phase.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment Group 1: Bictegravir (BIC)/ Lenacapavir (LEN) (75/50 mg) + PTM B/F/TAF (Experimental): Blinded Phase: Participants will switch from bictegravir/emtricitabine/tenofovir (B/F/TAF) FDC tablets to BIC/LEN (75/50 mg) FDC tablets and placebo-to-match (PTM) B/F/TAF. Participants will receive a 2-day oral loading dose of LEN 600 mg on Day 1 and on Day 2, in addition to the daily doses of BIC/LEN FDC tablet starting on Day 1 up to end of blinded treatment (EBT) visit.
  Open-label (OL) Phase: Following treatment in the Blinded Phase, participants from Treatment Group 1 will receive BIC/LEN FDC tablets through Week 48 in the Open-label Phase. At the OL Week 48 visit, participants from Treatment Group 1 will be given the option to continue to receive BIC/LEN FDC tablets until the conclusion of the OL Phase.
  Interventions: Drug: Bictegravir; Drug: Lenacapavir; Drug: Placebo to match B/F/TAF
- Treatment Group 2: B/F/TAF (50/200/25 mg) + PTM BIC/LEN (Experimental): Blinded Phase: Participants will continue with their B/F/TAF (50/200/25 mg) FDC tablets and start PTM BIC/LEN tablets on Day 1. Participants will receive PTM LEN tablets for 2 days (2 PTM LEN tablets on Day 1 and on Day 2. The blinded phase will continue until the EBT visit.
  Open Label Phase: Participants in Treatment Group 2 who complete the EBT visit will be given the option to enter the OL phase to receive BIC/LEN FDC tablets until the conclusion of the OL Phase.
  Interventions: Drug: Bictegravir; Drug: Lenacapavir; Drug: B/F/TAF; Drug: Placebo to match BIC/LEN

INTERVENTIONS:
Drug: Bictegravir — Tablets administered orally without regard to food
  Other Names: GS-9883
Drug: Lenacapavir — Tablets administered orally without regard to food
  Other Names: GS-6207
Drug: B/F/TAF — Tablets administered orally without regard to food
  Other Names: Biktarvy ®
  Arms: Treatment Group 2: B/F/TAF (50/200/25 mg) + PTM BIC/LEN
Drug: Placebo to match B/F/TAF — Tablets administered orally without regard to food
  Arms: Treatment Group 1: Bictegravir (BIC)/ Lenacapavir (LEN) (75/50 mg) + PTM B/F/TAF
Drug: Placebo to match BIC/LEN — Tablets administered orally without regard to food
  Arms: Treatment Group 2: B/F/TAF (50/200/25 mg) + PTM BIC/LEN

SUMMARY:
The goal of this clinical study is to learn more about the effects of switching to the study drugs, bictegravir (BIC)/lenacapavir (LEN), fixed-dose combination (FDC) versus current therapy bictegravir/emtricitabine/tenofovir alafenamide (B/F/TAF) FDC in people living with HIV-1 (PWH).

The primary objective of this study is to learn how effective it is to switch to BIC/LEN FDC tablets versus continuing on B/F/TAF FDC tablets in virologically suppressed PWH.

ELIGIBILITY:
Key Inclusion Criteria:

* Currently receiving B/F/TAF for at least 6 months prior to screening.
* If plasma human immunodeficiency virus type 1 (HIV-1) ribonucleic acid (RNA) measurements in the last 6 months prior to screening are available, all levels must be < 50 copies/mL.
* At least one documented HIV-1 RNA level measured between 6 and 12 months (± 2 months) prior to screening. This and any other HIV-1 RNA measurements documented in this period must be < 50 copies/mL.
* Plasma HIV-1 RNA levels < 50 copies/mL at screening.
* No documented or suspected resistance to BIC (including integrase strand-transfer inhibitor resistant (INSTI-R) mutations T66A/I/K, E92G/Q, G118R, F121Y, Y143C/H/R, S147G, Q148H/K/R, N155H/S, or R263K in the integrase gene).
* No documented or suspected resistance to tenofovir alafenamide (TAF) (TAF; mutations K65R, K65N, K70E, Q151M or T69 insertion, or ≥ 3 of the following thymidine analog mutations [M41L, D67N, K70R, L210W, T215Y/F, K219Q/E/N/R] in the reverse transcriptase gene).
* Estimated glomerular filtration rate ≥ 30 mL/min according to the Cockcroft-Gault formula for creatinine clearance.

Key Exclusion Criteria:

* Positive serum pregnancy test or pregnant at screening or a positive pregnancy test prior to Day 1 randomization.
* Breastfeeding (nursing).
* Prior use of, or exposure to, LEN.
* Active, serious infections (other than HIV-1) requiring parenteral therapy < 30 days prior to randomization.
* Active tuberculosis infection.
* Acute hepatitis < 30 days before randomization.
* Chronic hepatitis B virus (HBV) infection, as determined by either:

  * Positive HBV surface antigen and negative HBV surface antibody, regardless of HBV core antibody status, at the screening visit.
  * Positive HBV core antibody and negative HBV surface antibody, regardless of HBV surface antigen status, at the screening visit.
* Known hypersensitivity to the study drug, its metabolites, or any formulation excipient.
* History of or current clinical decompensated liver cirrhosis (eg, ascites, encephalopathy, or variceal bleeding).
* Abnormal electrocardiogram (ECG) at the screening visit that is clinically significant as determined by the investigator.
* Active malignancy requiring acute systemic therapy.
* Any of the following laboratory values at screening:

  * Alanine aminotransferase > 5 × upper limit of normal (ULN).
  * Direct bilirubin > 1.5 × ULN.
  * Platelets < 50,000/mm^3.
  * Hemoglobin < 8.0 g/dL.
* Requirement for ongoing therapy with or prior use of any prohibited medications listed in the protocol.
* Participation or planned participation in any other clinical study (including observational studies) without prior approval from the sponsor.
* Any other clinical condition or prior therapy that, in the opinion of the investigator, would make the participant unsuitable for the study or unable to comply with dosing requirements.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 577 (Actual)
Dates: Start 2024-03-25 (Actual); Primary Completion 2025-10-27 (Actual); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of Participants with HIV-1 RNA ≥ 50 copies/mL at Week 48 as Determined by the US FDA-defined Snapshot Algorithm | Week 48

SECONDARY OUTCOMES:
Proportion of Participants with HIV-1 RNA < 50 copies/mL at Week 48 as Determined by the US FDA-defined Snapshot Algorithm | Week 48
Change From Baseline in Clusters of Differentiation 4 (CD4) Cell Count at Week 48 | Baseline; Week 48
Treatment Group 1: Proportion of Participants with HIV-1 RNA ≥ 50 copies/mL at Week 96 as Determined by the US FDA-defined Snapshot Algorithm | Week 96
Treatment Group 1: Proportion of Participants with HIV-1 RNA < 50 copies/mL at Week 96 as Determined by US FDA-defined Snapshot Algorithm | Week 96
Treatment Group 1: Change from Baseline in CD4 Cell Count at Week 96 | Baseline; Week 96
Percentage of Participants Experiencing Treatment-Emergent Adverse Events (AEs) through Week 48 | From first dose date up to Week 48
Treatment Group 1: Percentage of Participants Experiencing Treatment-Emergent AEs through Week 96 | From first dose date up to Week 96

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (104):
- United States (51):
  - Pueblo Family Physicians, Phoenix, Arizona
  - Be Well Medical Center, Berkeley, California
  - Pacific Oaks Medical Group, Beverly Hills, California
  - Ruane Clinical Research Group Inc., Los Angeles, California
  - Alta Bates Summit Medical Center, Summit Campus, East Bay Advanced Care, Oakland, California
  - BIOS Clinical Research, Palm Springs, California
  - UCSD Anti Viral Research Centre (AVRC), San Diego, California
  - Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center, Torrance, California
  - Mills Clinical Research, West Hollywood, California
  - Public Health Institute at Denver Health, Denver, Colorado
  - Yale University School of Medicine (study visits), New Haven, Connecticut
  - Midland Florida Infectious Diseases Specialists, PL - Orange City, DeLand, Florida
  - Therafirst Medical Center, Fort Lauderdale, Florida
  - CAN Community Health, Fort Lauderdale, Florida
  - Midway Immunology and Research Center, Ft. Pierce, Florida
  - AIDS Healthcare Foundation - The Kinder Medical Group, Miami, Florida
  - Schiff Center for liver Diseases/University of Miami, Miami, Florida
  - Floridian Clinical Research, Miami Lakes, Florida
  - Orlando Immunology Center, Orlando, Florida
  - Bliss Healthcare, Orlando, Florida
  - AHF Pensacola, Pensacola, Florida
  - CAN community Health, Sarasota, Florida
  - Triple O Research Institute, P.A., West Palm Beach, Florida
  - Infectious Disease Specialists of Atlanta, Decatur, Georgia
  - Mercer University, Department of Internal Medicine, Macon, Georgia
  - Claudia T Martorell MD LLC dba The Research Institute, Springfield, Massachusetts
  - Henry Ford Health, Detroit, Michigan
  - KC Care health Center, Kansas City, Missouri
  - Southampton Community Healthcare, Inc., St Louis, Missouri
  - ID Care, LLC, Hillsborough, New Jersey
  - Saint Michael's Medical Center, Newark, New Jersey
  - New Jersey Medical School - Clinical Research Center, Newark, New Jersey
  - South Jersey Infectious Disease, Somers Point, New Jersey
  - AXCES Research Group, LLC, Santa Fe, New Mexico
  - New York-Presbyterian Queens, Flushing, New York
  - Montefiore Medical Center, The Bronx, New York
  - The Brody School of Medicine at East Carolina University , ECU Adult Specialty Care, Greenville, North Carolina
  - Rosedale Health and Wellness, Huntersville, North Carolina
  - Philadelphia FIGHT Community Health Centers, Philadelphia, Pennsylvania
  - Medical University of South Carolina (MUSC) Research Nexus, Charleston, South Carolina
  - Central Texas Clinical Research, Austin, Texas
  - St Hope Foundation, Inc., Bellaire, Texas
  - AIDS Arms, Inc. DBA Prism Health North Texas, Dallas, Texas
  - North Texas Infectious Diseases Consultants, PA, Dallas, Texas
  - AXCES Research Group, LLC, El Paso, Texas
  - Texas Centers for Infectious Disease Associates, Fort Worth, Texas
  - The Crofoot research Center, INC., Houston, Texas
  - AXCES Research Group, LLC, Salt Lake City, Utah
  - Clinical Alliance For Research & Education - Infectious Diseases. LLC (CARE-ID), Annandale, Virginia
  - Peter Shalit MD, Seattle, Washington
  - Community Health care, Tacoma, Washington
- Argentina (3):
  - Helios Salud S.A., Buenos Aires
  - Fundacion Huesped, Buenos Aires
  - Instituto CAICI SRL, Santa Fe
- Australia (3):
  - Taylor Square Private Clinic, Darlinghurst, New South Wales
  - Alfred Hospital(Alfred Health), Melbourne, Victoria
  - Prahran Market Clinic, South Yarra, Victoria
- Canada (6):
  - Chronic Viral Illness Service/McGill University Health Centre (MUHC), Decarie Montreal
  - Clinique Médicale l'Actuel, Montreal
  - The Ottawa Hospital - General Campus, Ottawa
  - Regina General Hospital, Regina
  - St. Paul's Hospital, John Ruedy Clinic-Immunodeficiency Clinic (JRC-IDC), Vancouver
  - Cool Aid Community Health Centre, Victoria
- Instituto Dominicano de Estudios Virologicos - IDEV, Santo Domingo, Dominican Republic
- Germany (7):
  - Praxis Dr. Knechten, Aachen
  - Novopraxis Berlin, Berlin
  - Praxis am Ebertplatz, Cologne
  - Universitätsklinikum Frankfurt, Frankfurt
  - Universitätsklinikum Hamburg Eppendorf, Hamburg
  - LMU Klinikum der Universität, Munich
  - Klinikum rechts der Isar der Technischen Universitaet Muenchen, München
- Italy (7):
  - ASST degli Spedali Civili di Brescia - Spedali Civili di Brescia - INCIPIT - PIN, Brescia
  - Azienda Ospedaliero Universitaria Ospedali Riuniti (Policlinico di Foggia), Foggia
  - IRCCS Ospedale San Raffaele, Milan
  - Fondazione IRCCS San Gerardo dei Tintori - ASST di Monza - A. O. San Gerardo, Monza
  - Fondazione IRCCS Policlinico San Matteo di Pavia, Pavia
  - Istituto Nazionale Malattie Infettive Lazzaro Spallanzani IRCCS, Roma
  - Fondazione Policlinico Universitario A Gemelli-Rome, Roma
- Japan (3):
  - National Hospital Organization Nagoya Medical Center, Aichi
  - National Hospital Organization Osaka National Hospital, Osaka
  - Center Hospital of the National Center for Global Health and Medicine, Tokyo
- Mexico (2):
  - ProcliniQ Investigacion Clinica Toriello Guerra, Tlalpan, Mexico City
  - Unidad de Atencion Medica e Investigacion en Salud, Mérida
- Puerto Rico (2):
  - HOPE Clinical Research, San Juan, PR
  - Proyecto ACTU, San Juan, PR
- South Korea (4):
  - Kyungpook National University Hospital, Daegu
  - National Medical Center, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul
- Spain (6):
  - Hospital Universitario Germans Trias i Pujol, Badalona Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Universitario La Paz - PPDS, Madrid
  - Hospital Universitario Virgen del Rocio - PPDS, Seville
  - Consorcio Hospital General Universitario de Valencia, Valencia
- Taiwan (4):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Kaohsiung Veterans General Hospital, Kaohsiung City
  - National Taiwan University Hospital, Taipei
  - Taoyuan General Hospital, Ministry of Health and Welfare, Taoyuan
- United Kingdom (5):
  - Liverpool University Hospitals NHS Foundation Trust, Royal Liverpool Hospital, Liverpool
  - King's College Hospital, Weston Education Centre, London
  - Chelsea and Westminster Hospital NHS Foundation Trust, St Stephen's Centre, Chelsea and Westminster Hospital, London
  - St Mary's Hospital - PPDS, London
  - Mortimer Market Centre, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Arora P, Hindman JT, West S, Ling J, Palaparthy R, Marathe DD. The effect of antacid and mineral supplements on bictegravir pharmacokinetics: results from a Phase 1, open-label, drug-drug interaction study. Antimicrob Agents Chemother. 2026 Jan 7;70(1):e0078125. doi: 10.1128/aac.00781-25. Epub 2025 Nov 28. PMID 41313173
- See also: Gilead Clinical Trials Website — https://www.gileadclinicaltrials.com/study?nctid=NCT06333808